CLINICAL TRIAL: NCT05037318
Title: From Threat to Challenge - Improving Medical Students' Stress Response and Communication Skills Performance Through the Combination of Stress Arousal Reappraisal and Preparatory Worked Example-based Learning When Breaking Bad News to Simulated Patients
Brief Title: Breaking Bad News - Optimizing Stress Response and Communication Performance in Medical Students
Acronym: BPSM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bern (Other)
Collaborators: Center for Primary Care and Public Health (Unisante), University of Lausanne, Switzerland (Other); University of Vienna (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Basic Science
Other Study IDs: BBN BPSM; 100019_200831 (Other Grant/Funding Number: Swiss National Science Foundation)
Record Dates: First submitted 2021-08-31; First posted 2021-09-08 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Stress Reaction
Keywords: Breaking bad news; Stress; Stress arousal reappraisal; Stressful communication; Communication skills; Worked example; Biopsychosocial model
MeSH Terms: conditions — Fractures, Stress

STUDY DESIGN:
Intervention Model Description: Two interventions are used, participants either receive only a stress reappraisal, only worked examples on breaking bad news, both interventions together, or none of the interventions.
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants know the content of their intervention, however, they do not know what other interventions there are and which group they belong to.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Stress arousal reappraisal (Experimental)
  Interventions: Behavioral: Stress arousal reappraisal
- Worked examples (Experimental)
  Interventions: Behavioral: Worked examples
- Stress arousal reappraisal + Worked examples (Experimental)
  Interventions: Behavioral: Stress arousal reappraisal; Behavioral: Worked examples
- Control (No Intervention)

INTERVENTIONS:
Behavioral: Stress arousal reappraisal — Participants will watch a video explaining that stress arousal is not harmful but rather functional and adaptive for performance in stressful situations.
  Arms: Stress arousal reappraisal; Stress arousal reappraisal + Worked examples
Behavioral: Worked examples — The worked example will be in form of brief video sequences showing a physician (played by an actor) delivering the bad diagnosis of lung cancer to an SP following the SPIKES protocol.
  Arms: Stress arousal reappraisal + Worked examples; Worked examples

SUMMARY:
Breaking bad news (e.g., telling patients that they have cancer) is not only very stressful for the patients concerned, but also for the physicians delivering the diagnosis. It is unclear how this burden and the associated communication performance can be optimized. The project contributes to this goal.

The main goal of the project is to scientifically analyze to what extent the stress reaction and communication performance of medical students can be optimized when breaking bad news. Two strategies will be employed and tested for their effectiveness: First, "stress arousal reappraisal", which consists in reinterpreting physiological arousal (e.g., increased heart rate) as adaptive and beneficial for task performance. Second, medical students can be well prepared for breaking bad news by learning from worked examples (step-by-step demonstrations of how to break bad news).

The investigators hypothesize that both strategies will shift the interpretation of breaking bad news from a threat to a challenge state. This will lead to better communication performance during the task.

To test the hypothesis, about 200 medical students' communication performance, cardiovascular activity, stress hormone release, and subjective stress perception when communicating a serious cancer diagnosis to a simulated patient (actor) will be measured.

The results of the study provide a first comprehensive picture of the psychophysiological stress patterns of medical students who are entrusted with a stressful communication task. Ultimately, this may promote stress management and communication skills in future physicians.

DETAILED DESCRIPTION:
Breaking bad news (BBN; e.g., telling patients that they have cancer) is a frequent task in the medical field. Appropriate communication when BBN is crucial for patient-related outcomes. For many physicians, BBN is a very demanding task often associated with high levels of stress, which can negatively impact their communication skills and health. It is thus important to provide future physicians with effective tools that enable them to cope successfully with their stress response and to perform the BBN task at their best. The planned project aims to contribute to this important goal in novel ways. One promising approach to improve people's stress response to demanding tasks is stress arousal reappraisal, which consists in reinterpreting physiological arousal as adaptive and beneficial for task performance. Recent work suggests that medical students can be well prepared for BBN by learning from worked examples (step-by-step demonstrations of how to break bad news).

Overall objectives: The study adopts the biopsychosocial model (BPSM) of challenge and threat as organizing theoretical framework to investigate the effects of stress arousal reappraisal and preparatory worked example-based BBN learning on the psychophysiological responses and communication skills performance of medical students tasked with BBN to simulated patients (SPs). The BPSM of challenge and threat holds that individuals are in a threat state when perceived resources fall short of perceived demands in a motivated performance situation, whereas they are in a challenge state when evaluated resources outweigh perceived demands. These states are primarily assessed with a self-reported resources-demands differential (perceived resources minus perceived demands) and a cardiovascular index (sum of cardiac output and reverse scored total peripheral resistance), with larger scores reflecting greater challenge. Secondarily, as suggested by recent research, they are also associated with salivary indices of the activity of the hypothalamic-pituitary-adrenal axis (cortisol and dehydroepiandrosterone) and of the sympatho-adrenal-medullary system (alpha-amylase). Compared to threats, challenge-type responses are associated with better task performance and better health outcomes.

Specific aims: The idea guiding the planned research is that both stress arousal reappraisal and preparatory worked example-based BBN learning will shift medical students' psychophysiological state from threat to challenge and by doing so their task performance will improve.

The hypotheses are: 1) students receiving stress arousal reappraisal instructions will show (i) more challenge-type psychophysiological responses and (ii) better BBN skills performance than students receiving no stress arousal reappraisal instructions; 2) students learning from a BBN-related worked example will show (iii) more challenge-type psychophysiological responses and (iv) better BBN skills performance than students not learning from a BBN-related worked example; 3) the challenge-threat resources-demands differential and cardiovascular index will be mediators of the effects of the interventions on BBN skills performance.

Method: A randomized controlled trial with a 2 (stress arousal reappraisal vs. no stress arousal reappraisal) x 2 (preparatory BBN learning with worked example vs. without worked example) between-subjects design with N = 200 Swiss medical students is envisioned. The investigators will assess participants' perceived task demands and coping resources, record their cardiovascular activity and collect their saliva before, during and after a videotaped BBN encounter with an SP. Three assessors will independently rate participants' BBN skills performance from the recordings.

Implications and relevance: Findings will support determining to what extent medical students' BBN-related stress responses and communication performance can be examined and understood from the challenge and threat perspective. Stress arousal reappraisal and preparatory worked example-based learning could be easily incorporated into the curriculum of medical students to help promote more adaptive challenge-type responses when facing BBN situations and potentially other stress-inducing communications with patients. This would ultimately have beneficial effects for both physicians and patients.

ELIGIBILITY:
Inclusion Criteria:

* Being currently enrolled as a third-year medical student
* Being German speaker
* Signed consent form

Exclusion Criteria:

* Cardiovascular diseases known to affect the variables under investigation
* Neuroendocrine conditions known to affect the variables under investigation
* Use of psychotropic drugs or any medication known to affect the variables under investigation (e.g., corticosteroids, cardioactive medication)
* Wearing a pacemaker
* Pregnancy/Breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 229 (Actual)
Dates: Start 2022-04-21 (Actual); Primary Completion 2024-02-29 (Actual); Study Completion 2024-02-29 (Actual)

PRIMARY OUTCOMES:
Breaking bad news performance | After 2 hours. Duration: 12 minutes
  SPIKES (6 items) and global Bad News Assessment Scale (glBAS; 5 items); both five-point ratings ranging from 1 to 5, glBAS is scored in reverse to match SPIKES scale, the higher the score, the better the performance

SECONDARY OUTCOMES:
Change in self-reported mood | During 3 hours, multiple pre and post intervention measures
  Multidimensional Mood State Questionnaire Short-scale; three dimensions, (8 items in total); 8-point scale; items have bipolar anchors (e.g., for valence, 1 = bad & 8 = good; calmness, 1 = tense, 8 = calm; energetic arousal, 1 = tired, 8 = awake)
Change in heart rate | During 3 hours, multiple pre and post intervention measures
  Heart beats per minute
Change in pre-ejection period | During 3 hours, multiple pre and post intervention measures
  Defined as the time in ms from the initiation of left-ventricle contraction to aortic-valve opening
Change in challenge-threat cardiovascular index | During 3 hours, multiple pre and post intervention measures
  Sum of cardiac output and reverse scored total peripheral resistance, z-Score
Change in anabolic balance | During 3 hours, multiple pre and post intervention measures
  Ratio of salivary cortisol to salivary dehydroepiandrosterone
Change in salivary alpha-amylase | During 3 hours, multiple pre and post intervention measures
  Concentration
Change in self-reported task resources-demands differential | 3 minutes before the intervention, 3 minutes before the BBN task, and 3 minutes after the BBN task
  2 items; "How demanding do you expect the task to be / was the task?", "How able are you / were you to cope with the demands of BBN task?"; 6-point Likert scale ranging from 1 "not at all" to 6 "extremely", score of first item is subtracted from the score of the second item, the higher the score, the more so is the task evaluated as a challenge, and less as a threat

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Berendonk, PD Dr., Principal Investigator — University of Bern
Locations (1):
- Institute for Medical Education, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication will be shared.
Time Frame: Data will be available as soon as the study is published.
Access Criteria: The investigators will make supplementary files and key datasets accompanying a publication to demonstrate reproducibility openly available in appropriate digital data repositories that conform to the Fair Data principles and maintained by a non-profit organisation. Specific datasets will be shared via domain-specific public repositories. Unstructured data will be shared via data repository Zenodo or Dryad. These data repositories fulfill biomedical journals' and SNSF's requirements (allowing publishing FAIR data, non-commercial).

REFERENCES:
- [Derived] Bosshard M, Schmitz FM, Guttormsen S, Nater UM, Gomez P, Berendonk C. From threat to challenge-Improving medical students' stress response and communication skills performance through the combination of stress arousal reappraisal and preparatory worked example-based learning when breaking bad news to simulated patients: study protocol for a randomized controlled trial. BMC Psychol. 2023 May 10;11(1):153. doi: 10.1186/s40359-023-01167-6. PMID 37165406